CLINICAL TRIAL: NCT00065559
Title: Treatment of Diabetic Nephropathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TRMTDN (terminated)
Record Dates: First submitted 2003-07-28; First posted 2003-07-31 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Celecoxib

INTERVENTIONS:
Drug: celecoxib

SUMMARY:
COX-2 is an enzyme that is found in several different tissues in the body. COX-2 appears to produce a substance called prostaglandins, mainly at sites of inflammation. Several drugs have been approved by the FDA that inhibit COX-2 such as celecoxib, or brand name Celebrex®. These drugs are primarily used in patients with osteoarthritis and rheumatoid arthritis to decrease inflammation and pain. COX-2 inhibitors have been developed because they are more selective in treatment of inflammation and pain and tend to have fewer gastrointestinal side effects than NSAIDs (nonsteroidal anti-inflammatory drugs) such as aspirin, ibuprofen, naproxen, etc.

The normal adult kidney expresses COX-2 in various regions. Prostaglandins, which are produced in the kidney by COX-2, may contribute to glomerular and tubulointerstitial inflammatory diseases (types of kidney diseases due to inflammation). In some animal studies, COX-2 inhibitors have been shown to be potentially beneficial in reducing the amount of protein spilled in the urine and preserving kidney function with these inflammatory kidney diseases. This study will compare the effects of COX-2 inhibitor to placebo (an inactive substance) in patients with diabetic nephropathy (kidney disease due to diabetes) and proteinuria (spilling protein in the urine) on 24-hour urinary protein excretion.

This study is designed to see whether COX-2 inhibitors are useful in treating diabetic patients with kidney disease. The purpose of this study is a short-term pilot study that will allow the gathering of important data such as the ability to carry out the study and carry it out safely. Subjects with proteinuria and diabetic kidney disease already on ACE (Angiotensin-Converting Enzyme) inhibitor or ARB (Angiotensin Receptor Blocker) therapy (types of blood pressure medicines) will be randomized to a type of study in which each subject will serve as their own control. The study is set up so that each subject will receive either the COX-2 inhibitor or placebo for a period followed by a period of no drug and then followed by a period of receiving either the COX-2 inhibitor or placebo (whichever they did not receive the first period).

DETAILED DESCRIPTION:
The study is designed with a screening period, a baseline period and a treatment period. The purpose of screening is to identify eligible subjects and to exclude ineligible subjects. A careful history and physical examination will be conducted to ensure that the subject meets all the inclusion criteria and does not meet any of the exclusion criteria. The screening period lasts from 2 days to 2 months in duration.

The baseline period is from 2 - 3 months in duration. During the first baseline visit, there is withdrawal of previously used angiotensin converting enzyme inhibitors or angiotensin receptor antagonists (if any) and the initiation of quinapril 20 mg daily therapy (or irbesartan --150 - 300 mg daily). The subject will then be seen as frequently as determined by the investigator for subject's safety. The purpose of the second baseline visit is to determine safety after the initiation of therapy quinapril 20 mg po per day (or irbesartan 150 - 300 mg per day). The purpose of third baseline visit is to insure that the subject meets all the inclusion and none of the exclusion criteria prior to randomization. In addition, it will be assured that the subject's blood pressure is at a safe level to proceed with randomization and the laboratory and urinary collections will be made.

Only those subjects who fulfill all inclusion and none of the exclusion criteria will proceed to randomization. Also, in order to proceed to the randomization phase of the study, the subject must have a blood pressure of less than or equal to 135/85mmHg.

The treatment phase will consist of 18 weeks. During the treatment phase, the subject will be followed for safety and efficacy. The subjects will be randomly assigned to COX-2 inhibitor for 6 weeks (1st 6 week cycle), washout 3 weeks, placebo 6 weeks (2nd 6 week cycle), washout 3 weeks or to placebo 6 weeks (1st 6 week cycle), washout 3 weeks, COX-2 inhibitor 6 weeks (2nd 6 week cycle), washout 3 weeks.

During baseline and treatment periods, interim visits will be held in order to address blood pressure control or other problems that the patient or the PI deems necessary for protocol adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Men or non-pregnant, non-lactating women with Type 1 or Type II diabetes and renal disease
* 24-hour urinary protein excretion greater than or equal to 500 mg
* Serum creatinine less than or equal to 3 mg/dl
* Willingness and ability to give informed consent and to cooperate with the protocol including discontinuing current antihypertensive medications if necessary

Exclusion Criteria:

* Pregnant or lactating women
* Renal disease other than diabetic nephropathy
* Renal Transplant or on dialysis
* Immunosuppressive agents for greater than 2 weeks in the 3 months prior to randomization (inhaled steroids are permissible)
* Renal vascular disease (uncorrected and hemodynamically significant)
* Obstructive uropathy (uncorrected and hemodynamically significant)
* History or evidence of acute renal failure within 6 months prior to randomization visit
* Serum potassium greater than 5.2 mEq/L
* Known human immunodeficiency virus disease (HIV)
* Any major disorder which in the opinion of the investigator would reduce life expectancy during the course of this study or could preclude participation in this or could adversely effect the interpretation of the data.
* Anticipated inability to cooperate with or any condition of sufficient severity to impair participation in the study.
* Any of the following cardiovascular conditions within 1 month of the screening visit: myocardial infarction, coronary angioplasty, coronary artery bypass graft, other revascularization procedure, severe or unstable angina, stroke, transient ischemic attack or hemodynamically important vascular disease.
* Need for chronic (greater than 2 weeks) immunosuppressive therapy including oral or IV corticosteroids. (Inhaled steroids are permissible.)
* History of drug sensitivity or adverse reaction to both ACE I and ARB.
* History of drug sensitivity, allergy, or adverse reaction to COX-2 inhibitor, aspirin, or sulfonamides.
* Evidence or suspicion of drug abuse or excessive alcohol consumption within 12 months prior to screening visit 1.
* Receipt of any investigational drug within 30 days or 5 half-lives of the investigational drug (the longer period will apply) before screening visit 1.
* Active psychiatric disorder.
* History of peptic ulcer disease and/or gastrointestinal bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-04; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rush Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Sinsakul M, Sika M, Rodby R, Middleton J, Shyr Y, Chen H, Han E, Lehrich R, Clyne S, Schulman G, Harris R, Lewis J. A randomized trial of a 6-week course of celecoxib on proteinuria in diabetic kidney disease. Am J Kidney Dis. 2007 Dec;50(6):946-51. doi: 10.1053/j.ajkd.2007.09.005. PMID 18037095